CLINICAL TRIAL: NCT02284360
Title: A Prospective Randomized Double-Blinded Placebo Controlled, Explorative Phase I Trial to Investigate the Safety and Tolerability of Two Different Doses of Topically Administered APOSEC™ in Healthy Male Subjects With Artificial Dermal Wounds
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Wolzt, Univ.-Prof. Dr.med.univ. Michael Wolzt, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MarsyasI
Record Dates: First submitted 2014-10-30; First posted 2014-11-06 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Healthy; Artificial Dermal Wound
Keywords: wound healing; APOSEC™; Safety
MeSH Terms: interventions — Administration, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Low dose (Experimental): Each volunteer in group A will receive both Verum and Placebo.
  The Verum lyophilized APOSEC™ is derived from 12.5*10^6 cells/ml irradiated lyophilized PBMC. The lyophilizate will be resuspended in 0.9% 200 µL NaCl and finally formulated in 800 µL Nugel.
  As Placebo a cell-free control lyophilisate resuspended in 0.9% 200 µL NaCl and finally formulated with 800 µL Nugel is used. The location of application on the inner upper arm (proximal or distal) of Verum and Placebo will be randomized.
  Interventions: Drug: APOSEC™ for cutaneous use
- Group B: High dose (Experimental): Each volunteer in group B will receive both Verum and Placebo.
  The Verum lyophilized APOSEC™ is derived from 25*10^6 cells/ml irradiated lyophilized PBMC. The lyophilizate will be resuspended in 0.9% 200 µL NaCl and finally formulated in 800 µL Nugel.
  As Placebo a cell-free control lyophilisate resuspended in 0.9% 200 µL NaCl and finally formulated with 800 µL Nugel is used. The location of application on the inner upper arm (proximal or distal) of Verum and Placebo will be randomized.
  Interventions: Drug: APOSEC™ for cutaneous use

INTERVENTIONS:
Drug: APOSEC™ for cutaneous use — On day 0, a blinded and randomized test treatment with Verum and Placebo is performed on intact skin. If the subject does not reveal any adverse events, the actual treatment phase is initiated 24h later.
  Following baseline evaluation on day 1, two punch biopsies (4mm) on the inner upper side of the non-dominant arm are set under local anesthesia. One wound on the upper arm (proximal or distal) will be treated with placebo and the second wound will be treated with the allocated concentration of Verum according to previous randomization scheme set for test treatment. Approximately 1ml of Verum vs. placebo will be applied on the artificial wounds.
  From day 2 to 6, artificial wounds will be cleaned with 0.9 % NaCl and then allocated treatment will be administered. Wound dressing will be done daily and will cover the whole area of application.
  On day 7 the treatment is terminated and the wound is evaluated with respect the extension of wound closure.

SUMMARY:
This is a prospective, single center, randomized, double-blinded, placebo-controlled, exploratory phase I clinical trial in healthy male subjects to investigate the safety and tolerability of the cytokine based gel APOSEC™. The proof of safety and tolerability of APOSEC™ is the primary objective. The secondary objective is to measure the extent of wound healing of APOSEC™.

DETAILED DESCRIPTION:
APOSEC™ is a human product derived from lyophilized conditional medium of peripheral blood mononuclear cells (PBMC) following 24 hours cultivation after irradiation with 60Gy. The soluble factors produced by these factors (secretome) have regenerative functions and enhance wound healing due to the activation of signaling cascades involved in the cell migration, proliferation and cell survival. The product also possesses strong angiogenic properties as well in vivo and in vitro. APOSEC™ is intended for topical use only, to promote healing of wounds in association with standard wound care. Standard wound care includes initial debridement, avoidance and treatment of wound related infections and a non-weight-bearing regime to decrease the pressure on the wound.

The verum APOSEC™ is processed as lyophilisate and resuspended in Nugel for the final formulation. It will be compared with a placebo, a cell-free parallel produced cell-free control lyophilisate that is finally formulated in Nugel as well.

10 eligible healthy volunteers will consecutively be allocated to 2 different dose groups of APOSEC™ in a dose escalation scheme. The first 5 subjects in group A receive the low dose of APOSEC™ (12.5*10^6 lyophilized PBMC/mL), the subsequent 5 subjects in group B will receive the high dose of APOSEC™ (25*10^6 lyophilized PBMC/mL). Each volunteer will receive both Verum and Placebo on two artificial wounds on the inner upper non-dominant arm. The location of application of the Verum and Placebo (proximal or distal) is subjected to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects with 18-50 years of age at the day of inclusion
* Written informed consent will be obtained prior to screening examination
* BMI of 19-27 (extremes included)
* Subjects are in good clinical and mental health as established by medical history, physical examination, vital signs, electrocardiogram, results of biochemistry, hematology, virology and urine analysis at the Screening Visit

Exclusion Criteria:

* Lack of willingness or capacity to co-operate appropriately
* Regular use of medications
* History of malignancies
* History of wound healing abnormalities
* Chronic dermatological disease
* History of chronic autoimmune diseases such as rheumatoid arthritis, inflammatory bowel disease, diabetes mellitus, Lupus erythematodus
* Tattoos in the region of planned punch biopsy
* Positive HIV serology or evidence of active hepatitis
* Allergy requiring medical treatment within 4 weeks before study initiation
* Active infection of fever > 38°C within 7 days prior randomisation
* Blood donation within 4 weeks before study initiation
* Clinically relevant abnormalities in the laboratory testing, vital signs, ECG or physical examination
* Participation in another clinical trial with an investigational day within 4 weeks before study participation

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
- The number of subjects experiencing Adverse Events, Serious Adverse Events, Dose-limiting toxicities or local tolerability issues as a measure of Safety and Tolerability will be assessed throughout the study period. | day 0 to day 17
  The primary objective is to investigate safety and tolerability of two different doses of APOSEC™ during the treatment and follow-up period of the study. Correspondingly, the primary endpoints are Adverse Events, Serious Adverse Events and Dose-limiting toxicities. Assessment of local tolerability or any adverse events will be accomplished by a score (expanding from no visible reaction to severe erythema with induration, vesicles / bullae / pustles / erosion / ulceration). Presence of local pain will be assessed by a Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
- Changes in wound size between baseline and End of Treatment (EOT) assessed by photographic analysis. | day 1 to day 7
  The secondary objectives are to investigate pharmacodynamic effects of APOSEC™ on wound healing during the treatment phase as well as on wound closure and scar formation after termination of the treatment, compared to placebo. Correspondingly the secondary endpoints are the change in wound size between baseline and end of treatment assessed by photographic analysis, that is retrospectively used for planimetric assessment. In addition to photographic analysis, the wound condition is evaluated with respect to its extension of re-epithelization / presence or absence of undermining and tunneling / presence of exsudate on the dressing.
Presence or absence of complete wound closure at End of Treatment (EOT) after Verum vs. Placebo administration. | day 7
  In terms of pharmacodynamic effects investigation, a further secondary endpoint is the presence of complete wound closure at end of treatment, which is assessed as dichotomic outcome.
- Scarring formation with respect to induration of palpable scar tissue. | day 7
  Evaluation of scar formation: The induraction of palpable scar tissue will be assessed in length and width [mm]. Moreover, the scar tissue will be evaluated using a caliper.
Presence or absence of re-epithelization and angiogenesis assessed by the markers CD31 and vWF. | day 1 / day 7
  The baseline biopsy specimen taken at day 1 prior initiation of treatment is histogically compared with the re-biopsy specimen taken on day 7 after termination of treatment.
  Baseline and re-biopsy specimens derived from randomized and blinded location of Verum application are compared to placebo. The biopsy specimens are histologically evaluated with respect to the extent of re-epithelization and angiogenesis by using CD31 and vWF as markers.
Investigator satisfaction assessment on applicability of the gel | day 0 - day 6
  Throughout the treatment period, the investigator shall evaluate the gel with respect to its applicability via a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria